CLINICAL TRIAL: NCT06713447
Title: A Pharmacokinetic Study of NTI164 in Healthy Adult Volunteers
Brief Title: NTI164 Human PK Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fenix Innovation Group (Industry)
Collaborators: CMAX Clinical Research Pty Ltd (Unknown); Neurotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FENPK1
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Healthy Volunteer
Keywords: Pharmacokinetic; Healthy; Cannabis
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Open-label, single intervention, single site pharmacokinetic study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NTI164 active (Experimental): All participants will be in this arm (single intervention) and will receive NTI164.
  Interventions: Drug: NTI164

INTERVENTIONS:
Drug: NTI164 — This intervention uses Full-Spectrum Medicinal Cannabis Plant Extract with a low THC concentration of 0.08% (NTI164) specifically formulated to target inflammation in various neurological conditions. The dose of 20mg/kg has been selected based off existing clinical trial evidence for NTI164, and is similar to the dose of other cannabis-based drugs used in neurology. The safety of NTI164 has been rigorously tested in several ongoing paediatric clinical trials through blood tests and clinician-rated surveys.

SUMMARY:
This study is looking at how a new cannabis compound with extremely low THC (0.08%), NTI164, is metabolised in the body and how it is excreted in urine over time (up to 28 days) in healthy adult volunteers. NTI164 will be delivered twice daily, at a concentration of 20mg/kg/day. There will be 2 parts to this study, Part A and Part B. Part A involves only one day of taking NTI164, whereas Part B involves taking NTI164 for 7 consecutive days. Urine samples and blood samples will be collected at certain time points after NTI164 dosing to help characterise how the drug is being broken down in the body and over what time frame.

DETAILED DESCRIPTION:
This open-label study aims to assess the efficacy of Full-Spectrum Medicinal Cannabis Plant Extract containing 0.08% THC (NTI164) in healthy adult volunteers. The main objective is to characterise the pharmacokinetic (PK) profile of NTI164 in the body. This study is split into 2 Parts, with NTI164 delivered orally twice daily at a dose of 20mg/kg/day (i.e. 2 x 10mg/kg doses), and blood and urine samples collected in both parts.

Part A involves only one day of NTI164 administration. In Part A, an oral dose of NTI164 will be administered to participants in a fasted state in the morning (AM). Blood samples will be collected at pre-dose and then 0.5, 2, 4, 6, and 8 hours following the AM dose. In the evening (PM), participants will receive another dose of NTI164 and bloods will be collected pre-PM dose, and 0.5, 2, 4, 6, 8, 12, and 24 hours following the PM dose.

On Day 3 and 4, only one blood sample will be collected in the morning. Urine samples will be collected pre-AM dose, as well as 4, 8, 12, and 24 hours following, and 4, 8, 16, and 24 hours following the PM dose. Following the 24-hour post-PM dose urine sample, urine samples will be collected every 6 hours until 72 hours after the initial AM dose on Day 1 (i.e. AM on Day 4).

Following blood and urine sample collection on Day 4, participants may be discharged from the clinical facility and will return on Day 7 to provide a final blood and urine sample. A follow-up phone call will be made to participants on Day 14 to ensure no adverse events have occurred and there are no concerns.

In Part B, NTI164 will be administered for 7 consecutive days. Participants will not need to be fasted for Part B. On Day 1 (day of first dose), blood samples will be collected at pre-dose and then 0.5, 2, 4, 6, and 8 hours following the AM dose. In the evening (PM), participants will receive another dose of NTI164, and bloods will be collected 0.5, 2, 4, 6, 8, 12, and 24 hours following the PM dose.

Urine samples will be collected pre-AM dose, as well as 4, 8, 12, and 24 hours following, and 4, 8, 16, and 24 hours following the PM dose. On Day 3, blood and urine samples will be collected pre-AM dose, and participants will be discharged and will continue at-home administration of NTI164.

Participants will return on Day 6 as intensive blood and urine sampling will occur once again on Day 7. On Day 7, blood samples will be collected at pre-dose and then 0.5, 2, 4, 6, 8, and 12 hours following the AM dose. In the evening (PM), participants will receive another dose of NTI164 (FINAL dose of the study), and bloods will be collected 0.5, 2, 4, and 24 hours (Day 8) following the PM dose. Urine samples will be collected pre-AM dose, as well as 4, 8, 12, and 24 hours following, and 4, 8, 16, and 24 hours following the PM dose.

The PM dose on Day 7 will be the final dose of NTI164 administered, however, participants will need to remain in the clinical facility on Day 8 for sample collection. A final blood and urine sample will be collected Day 9 AM, and then participants will be discharged from the clinical facility. Participants will return to the clinical facility for a blood and urine sample in the morning on Day 14, and also on Day 21 for a follow-up visit and final blood sample (no urine to be collected at this visit). This will mark the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are performed and must be able to understand the full nature and purpose of the study, including possible risks and AEs.
2. Adult males and females, 18 to 65 years of age (inclusive) at screening.
3. BMI ≥ 18.0 and ≤ 32.0 kg/m2, with a body weight of at least 50 kg.
4. Medically healthy (in the opinion of the Investigator), as determined by pre-study medical history and without clinically significant abnormalities. Must have:

   1. Physical examination without any clinically relevant findings;
   2. Systolic blood pressure (BP) in the range of 90 to 145 mmHg and diastolic BP in the range of 50 to 95 mmHg after resting for 5 minutes in a supine position.
   3. Pulse rate in the range of 45 to 100 bpm after 5 minutes resting in a supine position.
   4. Body temperature (tympanic), between 35.5°C and 37.7°C.
   5. Electrocardiogram (ECG) without clinically significant abnormalities including QT interval corrected for Fredericia (QTcF) <450 msec, QRS interval < 120 msec and PR interval < 220 msec, based on the average of triplicate measurements.
   6. No clinically significant findings in serum chemistry, haematology, coagulation, and urinalysis tests.
5. Female participants:

   1. Must be of non-child-bearing potential, i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 6 weeks before the screening visit or postmenopausal (with postmenopausal defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone (FSH) level consistent with postmenopausal status, per local laboratory guidelines), or
   2. If of child-bearing potential, must:

   i. Have a negative pregnancy test at the screening visit and on admission to the study site on Day-1. ii. Agree not to attempt to become pregnant or donate ova from signing the consent form until at least 30 days after the last dose of study drug. iii. Agree to use adequate contraception (defined as use of a condom by the male partner combined with use of a highly effective method of contraception (e.g. hormonal contraception, intrauterine device, bilateral tube occlusion, etc.) from one month prior to screening until at least 30 days after the last dose of study drug, if not exclusively in a same-sex relationship or abstinent as a committed lifestyle.
6. Male participants:

   1. Must agree not to donate sperm from signing the consent form until at least 90 days after the last dose of study drug.
   2. If engaging in sexual intercourse with a female partner who could become pregnant, agree to use adequate contraception (defined as use of a condom combined with use of a highly effective female method of contraception (as above)) from signing the consent form until at least 90 days after the last dose of study drug.
   3. If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, agree to use a condom from signing the consent form until at least 90 days after the last dose of study drug.
   4. Practise true abstinence: when this is in line with their preferred and usual lifestyle.
7. Have suitable venous access for blood sampling.
8. Abstain from alcohol for the duration of the study period.
9. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. Known hypersensitivity to any of the study drug ingredients.
2. History of anaphylaxis or other significant allergy (including system sensitivity to any aerosol) which, in the opinion of the Investigator, would interfere with the participant's ability to participate in the study.
3. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, psychiatric, or neurological disease/disorder, including any acute illness, determined by the Investigator to be clinically relevant.
4. Current diagnosis of bipolar disorder, major depressive disorder, psychosis, schizophrenia, or schizoaffective disorder.
5. History of major surgery or hospitalisation within 12 weeks prior to screening, or surgery planned during the study.
6. History of malignant disease in the last 10 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
7. Clinically relevant history or presence of rhythm disorders (e.g. sinoatrial heart block, second- or third-degree atrioventricular block, long QT syndrome, symptomatic bradycardia, atrial flutter, or atrial fibrillation), clinically-relevant history of hypokalaemia, congestive heart failure, or structural heart disease.
8. Presence or having sequelae of gastrointestinal, liver (with the exception of Gilbert's syndrome), kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
9. Serum or plasma potassium <3.5 or >5.2 mmol/L, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 x upper limit of normal (ULN), or total bilirubin >2 x ULN at screening or Day -1 (except for Gilbert's syndrome).
10. History of or positive test results for HIV, HBsAg, or HCV antibodies at screening.
11. Positive drugs of abuse test, urine cotinine test, and/or urine alcohol test results at screening and/or on admission to the clinical facility on Day -1.
12. History or clinical evidence of alcoholism or drug abuse (in the opinion of the Investigator) within the 3-year period prior to screening.
13. Regular consumption of >10 standard alcoholic beverages/week, where 1 standard drink is 10g of pure alcohol and is equivalent to 285 mL beer (4.9% Alc/Vol), 100 mL wine (12% Alc/Vol), or 30mL spirit (40% Alc/Vol).
14. Excessive caffeine consumption, defined as ≥ 800 mg per day at screening (1 cup of coffee contains ~100 mg caffeine, 1 cup of tea or one glass of cola contains ~40 mg caffeine, 1 can of Red Bull contains ~80 mg caffeine).
15. Females who are pregnant, breastfeeding, or planning to breastfeed.
16. Use of any prescribed medications (including vaccines) or over-the-counter medications (including herbal medicines, such as St John's Wort, homeopathic preparations, dietary supplements, vitamins, and minerals) within 2 weeks (or 5 half-lives, whichever is longer) prior to (first) study treatment administration, except the use of contraceptives, and occasional use of paracetamol and/or ibuprofen (at the discretion of the Investigator).
17. Received any vaccinations within 14 days prior to screening.
18. Donation of blood or plasma within 12 weeks prior to screening, loss of whole blood of >500mL within 12 weeks prior to first dose of study drug, or receipt of a blood transfusion within 1 year of first dose of study drug.
19. Participation in another clinical study of an investigational drug or device within 12 weeks prior to screening.
20. Any other condition or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.
21. Currently using or has used recreational or medicinal cannabis or cannabinoid-based medications within the 12 weeks prior to screening and is unwilling to abstain for the duration of the study.
22. Had brain surgery or a traumatic brain injury within 1 year of screening.
23. History of suicidal behaviour or suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the 12 weeks prior to screening and in ongoing assessment throughout the study.
24. Has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | Up to 21 days
  Maximum concentration of the drug at timepoints: baseline (pre-dose), 1, 2, 3, 4, 5, 12, 24 hrs post commencement of treatment, and daily up to 7 days post-dose for Part A and 21 days for Part B.

SECONDARY OUTCOMES:
Ae t1-t2 - urine | Up to 21 days
  Amount of drug excreted in urine at timepoints: baseline (pre-dose), 1, 2, 3, 4, 5, 12, 24 hrs post commencement of treatment, and daily up to 7 days post-dose for Part A and 21 days for Part B.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as per commercial in confidence restrictions.